CLINICAL TRIAL: NCT03496740
Title: Ultrasound Guided Dorsal Penile Block vs Neurostimulator Guided Pudendal Block in Children Undergoing Hypospadias Surgery: A Prospective, Randomized, Double-Blind Trial
Brief Title: Ultrasound Guided Penile Block vs Pudendal Block for Hypospadias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-379
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Ultrasound; Dorsal Penile Nerve Block; Pudendal Block; Hypospadias
MeSH Terms: conditions — Pain, Postoperative; Hypospadias | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penile Block (Active Comparator): Ultrasound guided dorsal penile nerve block will be administered after general anesthesia.
  0,25% Bupivacaine 0,5ml/kg (max. 20ml) will be used for the blocks
  Interventions: Procedure: Penile Block; Drug: Bupivacaine (Block Drug)
- Pudendal Block (Active Comparator): Nerve stimulator-guided pudendal block. 0,25% Bupivacaine 0,5ml/kg (max. 20ml) will be used for the blocks
  Interventions: Procedure: Pudendal Block; Drug: Bupivacaine (Block Drug)

INTERVENTIONS:
Procedure: Penile Block — Ultrasound guided dorsal penile nerve block will be done to this group of patients preoperatively, under general anesthesia. 0,25% Bupivacaine 0,5ml/kg (max. 20ml)
  Arms: Penile Block
Procedure: Pudendal Block — Nerve stimulation guided bilateral pudendal block will be done to this group of patients preoperatively, under general anesthesia. 0,25% Bupivacaine 0,5ml/kg (max. 20ml)
  Arms: Pudendal Block
Drug: Bupivacaine (Block Drug) — Block drug

SUMMARY:
Pain after hypospadias surgery is a challenging issue to solve for anesthesists. Many different analgesia techniques were defined in literature for this purpose. The investigators have implemented application of ultrasound guided dorsal penile nerve block into practice for these type of surgeries. Main purpose of this study is to compare the efficacy of nerve stimulator guided pudendal nerve block with ultrasound guided dorsal penile nerve block for postoperative analgesia after hypospadias surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1 to 10 years of age
* ASA I-II
* Undergoing elective hypospadias surgery

Exclusion Criteria:

* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* ASA III-IV
* Patients with neurological disorders

Ages: 1 Year to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male patients undergoing elective hypospadias surgery
Enrollment: 36 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic | postoperative 7 day
  First need for rescue analgesic after the surgery will be recorded

SECONDARY OUTCOMES:
Pain Scores | postoperative 48 hour
  FLACC scale will be used. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided